CLINICAL TRIAL: NCT02115243
Title: A Phase I Trial of Neoadjuvant Ipilimumab Followed by Melphalan Via Isolated Limb Infusion for Patients With Unresectable In-transit Extremity Melanoma
Brief Title: Trial of Neoadjuvant Ipilimumab Followed by Melphalan Via Isolated Limb Infusion for Patients With Unresectable In-transit Extremity Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00046479
Record Dates: First submitted 2014-04-12; First posted 2014-04-15 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Unresectable Melanoma
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipi/ILI (Other): Patients will receive ipilimumab followed by ILI.
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab

SUMMARY:
The purpose of this study is to determine safety profile, initial response rates and progression free survival for the combination therapy of neoadjuvant system ipilimumab followed by ILI with melphalan in patients with in transit melanoma.

Hypothesis:

The combination of regional LPAm plus systemic ipilimumab will lead to a larger response rate than either therapy alone.

The combination of regional LPAm plus systemic ipilimumab will cause larger changes in immune cell populations than are seen with either therapy along.

Changes in immune cell populations will predict progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically proven primary or recurrent extremity melanoma, stage IIIB, IIIC, or stage IV (AJCC staging must be documented in patient's medical record, as determined by CT of the chest, abdomen and pelvis, and/or whole body PET scan, and MRI of the brain within 4 weeks prior to administration of study drug)
2. Patients with Stage IV disease must have had all distant disease resected at least 30 days prior to regional treatment.
3. Patient must be greater than 18 years of age.
4. Patient must have an ECOG/Zubrod status of 0-1.
5. Patient's disease must be bi-dimensionally measurable by caliper or radiological method as defined in the RECIST criteria. For subjects with a single lesion, archived tissue must be available for research analysis. The sum of target lesion diameters should be at least 10 mm.
6. Disease to be treated by ILI must be distal to the planned site of tourniquet placement (which for the leg is generally the apex of the femoral triangle, or for the arm is distal to the deltoid insertion). If provider feels ILI appropriate with disease in these areas, patient may be enrolled with PI approval.
7. Patient must have adequate bone marrow, liver and renal function as assessed by the following:

   1. Hemoglobin greater than 9.0 g/dl
   2. White blood count (WBC) of greater than 2000 m3
   3. Absolute neutrophil count (ANC) greater than 1,000/mm3
   4. Platelet count greater than 75,000/mm3
   5. Total bilirubin less than 2.0 x ULN
   6. ALT and AST less than 2.5 x the ULN
   7. Creatinine less than 2.0 x ULN
8. Patient must have a palpable femoral/radial pulse in the affected extremity.
9. Patients must have a life expectancy of greater than 6 months.
10. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

    1. Amenorrhea greater than 12 consecutive months without another cause, or
    2. For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level greater than 35 mIU/mL.

    Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

    WOCBP must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.

    Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
11. Patient must provide a signed and dated written informed consent prior to registration and any study-related procedures.
12. Patient must provide written authorization to allow the use and disclosure of their protected health information at any institution subject to US HIPAA regulations.
13. Ability to read and understand English and the ability to complete paper +/- electronic survey assessments.

Exclusion Criteria:

1. Cardiac disease: Congestive heart failure greater than class II NYHA. Patients must not have unstable angina (angina symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
2. Autoimmune disease: History of or current active autoimmune diseases, [e.g. including but not limited to inflammatory bowel diseases [IBD], rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barre syndrome). Vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are not exclusionary.]
3. Prior allogeneic stem cell transplantation.
4. Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
5. History of or current immunodeficiency disease [e.g. splenectomy or splenic irradiation].
6. Psychiatric conditions or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance; any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
7. Concomitant therapy with any of the following: IL 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses). However, during the course of the study, use of corticosteroids is allowed if used for treating irAEs, adrenal insufficiencies, or if administered at doses of prednisone greater than or equal to 7.5mg daily or equivalent.
8. Women of childbearing potential (WOCBP), defined above in Section 5.1, who:

   1. are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug, or
   2. have a positive pregnancy test at baseline, or
   3. are pregnant or breastfeeding.
9. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 26 weeks after ipilimumab is stopped.

   Sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test before first receiving ipilimumab. If the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study.
10. Known brain metastasis.
11. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
12. Active clinically serious infection greater than CTCAE Grade 2.
13. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
14. Pulmonary hemorrhage/bleeding event greater than CTCAE Grade 2 within 4 weeks of study entry.
15. Any other hemorrhage/bleeding event greater than CTCAE Grade 3 within 4 weeks of study entry.
16. Evidence or history of bleeding diathesis or coagulopathy.
17. Antineoplastic therapy, radiotherapy, or any other investigational drug within 30 days prior to first study drug administration.
18. Current treatment, or treatment in the previous 24 months, for another non-melanoma malignancy, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the cervix.
19. Unable to return at the regular required intervals for reassessment, or study drug administration.
20. Patients with known heparin induced thrombocytopenia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 2 years
  The primary objective is to characterize the safety and tolerability of combining IPI and ILI by determining the MTD of IPI when used prior to ILI with LPAM.

SECONDARY OUTCOMES:
Response Rate | 3 years
  Estimate the complete response rate to ipi plus ILI in the patients who received the MTD of ipi.
Progression Free Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Tyler, MD, Principal Investigator — Duke University; April K Salama, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States